CLINICAL TRIAL: NCT03493932
Title: Cytokine Microdialysis For Real Time Immune Monitoring in Glioblastoma Patients Undergoing Checkpoint Blockade
Brief Title: Cytokine Microdialysis for Real-Time Immune Monitoring in Glioblastoma Patients Undergoing Checkpoint Blockade
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180077; 18-N-0077
Record Dates: First submitted 2018-04-10; First posted 2018-04-11 (Actual); Results first posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2023-09

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Glioma; Brain Tumor; Immune Therapy; Checkpoint Inhibition
MeSH Terms: conditions — Glioblastoma; Glioma; Brain Neoplasms | interventions — Nivolumab; relatlimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab and BMS-986016 (Experimental): Recurrent Glioblastoma patients
  Interventions: Drug: Nivolumab; Drug: BMS-986016

INTERVENTIONS:
Drug: Nivolumab — OPDIVO is a human programmed death receptor-1 (PD-1) blocking antibody indicated for the treatment of patients with unresectable or metastatic melanoma and disease progression following ipilimumab and, if BRAF V600 mutation positive, a BRAF inhibitor.
Drug: BMS-986016 — Anti-Lymphocyte Activation Gene-3 antibody undergoing clinical evaluation by Bristol-Myers Squibb

SUMMARY:
Background:

Glioblastoma (GBM) brain tumors almost always return after treatment. When that happens the tumor can never completely be removed by surgery, so most people also receive drugs. Researchers want to see if combining the drugs nivolumab and BMS-986016 may help.

Objectives:

To study how nivolumab affects the brain s immune system in people who have had glioblastoma brain tumors return. To study how nivolumab and BMS-986016 affect brain tumors.

Eligibility:

Adults age 18 and older who have had a return of GBM

Design:

Participants will be screened with:

Medical history

Physical exam

Cheek swab

Heart, blood and urine tests

Chest x-ray

Magnetic resonance imaging (MRI) brain scan. Participants will lie on a table that slides in and out of a cylinder in a strong magnetic field. A contrast agent will be injected in an arm vein.

Participants will stay in the hospital. They will:

Have surgery. A tube will be inserted into the back. Brain tumor and bone marrow samples will be taken. Tubes will be inserted into the brain.

Have a computed tomography brain scan.

Stay in Intensive Care (ICU) 7 days. Fluid from the brain and back will be collected every few hours. In the ICU, participants will get nivolumab by IV for 30 minutes.

Have surgery to remove the tubes.

Have standard surgery to remove as much of the GBM as possible. Bone marrow will be removed.

After leaving the hospital, participants will have visits every 2 weeks to get the study drugs by IV and have physical exams and blood tests.

Participants will have a brain MRI once a month.

...

DETAILED DESCRIPTION:
Objective

This protocol is being performed to 1) characterize the clinical and 2) immunological response of patients with recurrent glioblastoma to treatment with Nivolumab, together with an anti-Lag-3 antibody, BMS-986016, and to evaluate the safety of brain tumor microdialysis in this patient population.

Study Population

10 patients (total, after replacement for any dropout), 18 years old and older with recurrence of glioblastoma after standard treatment of surgery, chemotherapy, and radiation.

Study Design

Patients will be screened by study neurosurgeons or neuro-oncologists to verify their confirmed or likely diagnosis of a recurrent glioblastoma. Patients will be offered standard of care therapy, including repeat surgery and/or recommendations for chemotherapeutic agents and other trials. If the patients are deemed to be surgical candidates for their potential recurrence, they will be enrolled in the trial. Enrolled patients will then undergo a stereotactic brain biopsy. If a frozen section confirms a diagnosis of recurrent glioblastoma, two microdialysis catheters will be placed in the brain after the biopsy, and a lumbar drain will also be placed. These microdialysis catheters will sample interstitial fluid in and around the brain tumor every 6 hours. We will collect blood and cerebral spinal fluid samples daily for comparison. After two days (Day 3), the patients will be given one dose of Nivolumab, 240mg IV. We will continue to collect samples every six hours from the microdialysis catheters and daily from blood and cerebral spinal fluid for 5 additional days, after which patients will undergo surgical resection of their tumors and removal of the microdialysis catheters and lumbar drain. Nivolumab, at a dose of 240mg IV over 30 minutes every 2 weeks, will be administered after surgery (starting on Day 17(+/- 2 days), two weeks after the first dose on Day 3) followed by BMS 986016, an anti-Lag-3 antibody at a dose of 80mg IV over 60 minutes, until the study neuroradiologist notes tumor progression on MRI or the patient experiences treatment toxicity. While on therapy with Nivolumab and BMS-986016, patients will be seen and examined every 2 weeks +/- two days for signs of toxicity. Patients will be followed for at least three months after the surgical procedure.

Outcome Measures

The primary outcome measures are the proportion of patients who have a measurable increase of interferon gamma levels in the brain tumor tissue after their first dose of Nivolumab as compared to the pre-treatment baseline, the safety of using brain tumor microdialysis to monitor response to immune modulators in patients with recurrent glioblastoma and the safety of the combination of Nivolumab and BMS-986016. Exploratory outcome measures include: 1) To determine the change in interferon gamma production within the tumor microenvironment and in the rest of the body from before and after therapy with the immune checkpoint inhibitor, nivolumab; 2) To evaluate the pathological response of the immune microenvironment of brain tumor tissue to the first dose of Nivolumab; 3) To evaluate the clinical response (progression free survival, overall survival) of recurrent glioblastoma patients to this treatment combination; 4) To describe the difference in survival between responders and non-responders on this treatment combination; 5) To examine the differences in the immune cells and secreted factors of the tumor environment as compared to the immune cells and secreted factors of the cerebral spinal fluid, blood and, potentially, bone marrow in response to this treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for entry into the study, a candidate must meet all the following criteria:

1. Be 18 years of age or older.
2. Have recurrent glioblastoma that is amenable to surgical resection.
3. Agree to undergo brain surgery.
4. Are eligible for 03-N-0164 "Evaluation and Treatment of Neurosurgical Disorders" protocol 5. Willing and able to appoint a durable power of attorney.
5. Willing and able to appoint a durable power of attorney
6. Are willing to use an effective method of contraception during the clinical study as defined on the consent and for 24 weeks (for women) or 33 weeks (for men) after the last dose of the study drug.

EXCLUSION CRITERIA:

Candidates will be excluded if they:

1. Have a bleeding disorder that cannot be corrected before invasive testing or surgery, or other medical conditions that would make surgery unsafe, such as lung or cardiac disease that would render them unable to tolerate the risk of general anesthesia, or severe immunodeficiency.
2. Has a known additional malignancy that is progressing or requires active treatment within 3 years of registration. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
3. Are pregnant or breastfeeding
4. Cannot have an MRI scan.
5. Are claustrophobic
6. Are not able to lie on their back for up to 60 minutes
7. Have primary CNS lymphoma.
8. Has received systemic immunosuppressive treatments, aside from systemic corticosteroids (such as methotrexate, chloroquine, azathioprine, etc) within six months of registration
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
10. Have a significant cardiac history, such as 2 or more MIs OR 2 or more coronary revascularization procedures.
11. Have abnormal findings on ECG such as prolonged QT interval, T-wave abnormalities or arrhythmia. Abnormal findings on ECG will prompt an evaluation by a cardiologist prior to enrollment in the study
12. Are currently undergoing treatment with another therapeutic agent for glioblastoma
13. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti- Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
14. Have an ejection fraction less than 50% on screening echocardiogram
15. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies) at the time of enrollment
16. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected) at the time of enrollment.
17. Have an active infection that requires systemic antibacterial, antiviral or antifungal therapy Less than 7 days prior to initiation of study drug therapy
18. Have a history of transfer of autologous or allogeneic T cells
19. Have a history of solid organ or tissue transplants
20. Have cardiac Troponin T or I greater than 2 times the institutional upper limit of normal at screening
21. At the time of enrollment, lack of consent capacity due to cognitive impairment that would make them incapable of understanding the explanation of the procedures in this study. Cognitive capacity to consent will be determined at the time of enrollment. Patients with mental disorders or those patients who are cognitively impaired yet still retain consent capacity will not be excluded.
22. Cannot speak English or Spanish fluently
23. Patients that require dexamethasone greater than 4 mg/ day or equivalent of steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sadhana Jackson, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - National Institutes of Health Clinical Center, Bethesda, Maryland

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-N-0077.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Nivolumab and BMS-986016: Nivolumab: OPDIVO is a human programmed death receptor-1 (PD-1) blocking antibody indicated for the treatment of patients with unresectable or metastatic melanoma and disease progression following ipilimumab and, if BRAF V600 mutation positive, a BRAF inhibitor.
  BMS-986016: Anti-Lymphocyte Activation Gene-3 antibody undergoing clinical evaluation by Bristol-Myers Squibb
Period: Overall Study
Arm/Group | Experimental: Nivolumab and BMS-986016
Started | 21
Completed | 13
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: Nivolumab and BMS-986016
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Increase of Interferon Gamma Levels
Description: The proportion of patients that have a rise in interferon gamma levels within the tumor microenvironment of 4 pg/ml or higher before the first dose of Nivolumab as compared to the 5th day after treatment with Nivolumab.
Time Frame: Day 8
Measure: Count of Participants; unit: Participants
Groups:
- Recurrent Glioblastoma Patients: Nivolumab: OPDIVO is a human programmed death receptor-1 (PD-1) blocking antibody indicated for the treatment of patients with unresectable or metastatic melanoma and disease progression following ipilimumab and, if BRAF V600 mutation positive, a BRAF inhibitor.
  BMS-986016: Anti-Lymphocyte Activation Gene-3 antibody undergoing clinical evaluation by Bristol-Myers Squibb
Arm/Group | Recurrent Glioblastoma Patients
Number analyzed (Participants) | 13
Participants | 0

2. Primary Outcome: Microdialysis Catheter
Description: The number of patients with any adverse events that are directly attributable to placement of the microdialysis catheter. Specifically, intracranial hemorrhage, intracranial infection, wound infection, or new neurological deficit attributable to location of microdialysis catheter placement were to be captured
Time Frame: Day 8
Measure: Count of Participants; unit: Participants
Arm/Group | Recurrent Glioblastoma Patients
Number analyzed (Participants) | 13
Participants | 13

3. Primary Outcome: Drug Safety
Description: The safety of the combination of nivolumab and BMS-986016 in recurrent glioblastoma patients
Time Frame: Day 8
Measure: Number; unit: events attributed to nivolumab/BMS-98601
Arm/Group | Nivolumab and BMS-986016
Number analyzed (Participants) | 13
events attributed to nivolumab/BMS-98601 | 117

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Recurrent Glioblastoma Patients
All-Cause Mortality (participants affected / at risk) | 13/13
Serious Adverse Events (participants affected / at risk) | 13/13
Other Adverse Events (participants affected / at risk) | 1/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recurrent Glioblastoma Patients (N=13)
Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Recurrent Glioblastoma Patients (N=13)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1
White blood cell decreased (Blood and lymphatic system disorders) | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1
Neutrophil count decreased (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Elevated WBC count (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
ALC low (Blood and lymphatic system disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Hyperglycemia (Endocrine disorders) | 1
Abnormal thyroid function tests (Endocrine disorders) | 1
Cushingoid (Endocrine disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Alkalosis (Metabolism and nutrition disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Investigations - Other specify (Investigations) | 1
GGT increased (Investigations) | 1
CK increased (Investigations) | 1
elevated total bilirubin (Investigations) | 1
elevated AST (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 1
Fever (General disorders) | 1
Fatigue (General disorders) | 1
Chills (General disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Fecal incontinence (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Anorectal infection (Gastrointestinal disorders) | 1
Blurred Vision (Eye disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
atrial fibrillation (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 1
Li Fraumeni Syndrome (Congenital, familial and genetic disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Wound dehisence of biopsy site (Injury, poisoning and procedural complications) | 1
extremity weakness (Musculoskeletal and connective tissue disorders) | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Insomnia (Psychiatric disorders) | 1
Urinary Incontinence (Renal and urinary disorders) | 1
urinary urgency (Renal and urinary disorders) | 1
benign prostate hypertrophy (Reproductive system and breast disorders) | 1
Flushing (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify - limited skin erythema only, asymptomatic (Skin and subcutaneous tissue disorders) | 1
pruritis (Skin and subcutaneous tissue disorders) | 1
Petechial rash (Skin and subcutaneous tissue disorders) | 1
Macular rash (Skin and subcutaneous tissue disorders) | 1
Papular erythematous rash on upper extremities (Skin and subcutaneous tissue disorders) | 1
Folliculitis (Skin and subcutaneous tissue disorders) | 1
rash (Skin and subcutaneous tissue disorders) | 1
Pityrosporum folliculitis (Skin and subcutaneous tissue disorders) | 1
sweating (Skin and subcutaneous tissue disorders) | 1
sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
balance instability (Nervous system disorders) | 1
Cerebral edema (Nervous system disorders) | 1
change with cognition "fuzzy cognition (Nervous system disorders) | 1
Communicating hydrocephalus (Nervous system disorders) | 1
Difficulty reading (Nervous system disorders) | 1
Drowsiness (Nervous system disorders) | 1
dysphasia (Nervous system disorders) | 1
Edema, cerebral (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
intracranial edema (Nervous system disorders) | 1
Intracranial Hemorrhage (CT) (Nervous system disorders) | 1
Left facial droop (Nervous system disorders) | 1
left facial weakness (Nervous system disorders) | 1
left hemiparesis (Nervous system disorders) | 1
Left lower quadrantanopsia (Nervous system disorders) | 1
Left superior quadrantanopsia (Nervous system disorders) | 1
Mental Fogginess- distraction (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Photophobia (Nervous system disorders) | 1
Positive pronator drift test (Nervous system disorders) | 1
Pre-syncope (Nervous system disorders) | 1
Facial muscle weakness (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Short term memory difficulty (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Stroke (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT03493932/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/32/NCT03493932/ICF_001.pdf